CLINICAL TRIAL: NCT01508923
Title: Effect of NNC 90-1170 on 24-hour Glucose and Hormonal Profiles, Gastric Emptying, and Fasting Gluconeogenesis in Type 2 Diabetic Subjects. A Double-blind, Placebo-controlled, Randomised, Cross-over Trial
Brief Title: Effect of Liraglutide on Glucose Profiles and Gastric Emptying in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-1332
Record Dates: First submitted 2012-01-09; First posted 2012-01-12 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment period 1 (Experimental)
  Interventions: Drug: liraglutide; Drug: placebo
- Treatment period 2 (Placebo Comparator)
  Interventions: Drug: liraglutide; Drug: placebo

INTERVENTIONS:
Drug: liraglutide — 6 mcg/kg injected subcutaneously daily in each treatment period in random order. In total, subjects are treated 9-10 days
  Other Names: NNC 90-1170
Drug: placebo — 6 mcg/kg injected subcutaneously daily in each treatment period in random order. In total, subjects are treated 9-10 days

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to determine the effect of NNC 90-1170 (liraglutide) on glucose and hormonal profiles, fasting gluconeogenesis and insulin secretion in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Diet treated and/or subjects in monotherapy with max. 50 % of maximal dose of sulphonylurea (SU). In addition, subjects in treatment with metformin and/or repaglinide could be included
* Body Mass Index (BMI) maximum 35 kg/m^2
* Fasting plasma glucose 7-15 mmol/l, both inclusive

Exclusion Criteria:

* Impaired liver function
* Impaired renal function
* Anaemia
* Cardiac disease
* Uncontrolled treated/untreated hypertension
* Recurrent major hypoglycaemia as judged by the Investigator
* Known or suspected allergy to trial product or related products
* Females of child bearing potential who are pregnant, breast-feeding or have intention of becoming pregnant or are not using adequate contraceptive measures
* Current treatment with thiazolidinediones or chronic daily use of insulin (more than 7 days) within three months in the absence of intercurrent illness
* Loss of more than 400 ml blood during the three months prior to study start
* Allergy to paracetamol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2001-05; Primary Completion 2002-02 (Actual); Study Completion 2002-02 (Actual)

PRIMARY OUTCOMES:
24-hour glucose profiles after three fixed meals

SECONDARY OUTCOMES:
24-hour insulin profiles after three fixed meals
First phase insulin and maximal insulin secretory capacity
EGR (endogenous glucose release) expressed in mg/kg/min
GNG (gluconeogenesis) expressed in mg/kg/min
24-hour glucagon profiles after three fixed meals
24-hour FFA (free fatty acids) profiles after three fixed meals
4-hour paracetamol profiles after two fixed meals
30-hour NNC 90-1170 profile
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Århus C, Denmark

REFERENCES:
- [Result] Degn KB, Juhl CB, Sturis J, Jakobsen G, Brock B, Chandramouli V, Rungby J, Landau BR, Schmitz O. One week's treatment with the long-acting glucagon-like peptide 1 derivative liraglutide (NN2211) markedly improves 24-h glycemia and alpha- and beta-cell function and reduces endogenous glucose release in patients with type 2 diabetes. Diabetes. 2004 May;53(5):1187-94. doi: 10.2337/diabetes.53.5.1187. PMID 15111485
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com